CLINICAL TRIAL: NCT01086540
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II Multicenter Trial of a Monoclonal Antibody to CD20 (Rituximab) for the Treatment of Systemic Sclerosis-Associated Pulmonary Arterial Hypertension (SSc-PAH)
Brief Title: Rituximab for Treatment of Systemic Sclerosis-Associated Pulmonary Arterial Hypertension (SSc-PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ASC01
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Systemic Sclerosis-Associated PAH
Keywords: Pulmonary Arterial Hypertension (PAH); Autoimmune Disease; Systemic Scleroderma
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Autoimmune Diseases; Scleroderma, Systemic | interventions — Rituximab; Prednisone; Methylprednisolone; Adrenal Cortex Hormones; Diphenhydramine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab+PAH SOC (Experimental): Rituximab (1000 mg) will be administered as 2 intravenous infusions given 2 weeks apart.
  Concurrent stable-dose Pulmonary Arterial Hypertension (PAH) medical therapy will be continued/managed as per standard of care (PAH SOC).
  Interventions: Biological: Rituximab; Diagnostic Test: CMRI; Drug: prednisone; Drug: methylprednisolone; Drug: diphenhydramine; Drug: acetaminophen
- Placebo + PAH SOC (Placebo Comparator): Placebo will be administered as 2 intravenous infusions given 2 weeks apart.
  Concurrent stable-dose Pulmonary Arterial Hypertension (PAH) medical therapy will be continued/managed as per standard of care (PAH SOC).
  Interventions: Other: Placebo; Diagnostic Test: CMRI; Drug: prednisone; Drug: methylprednisolone; Drug: diphenhydramine; Drug: acetaminophen

INTERVENTIONS:
Biological: Rituximab — Participants receive rituximab intravenous (IV) infusions, 1000 mg each, 14 days apart (Day 0 and Week 2).
  Rituximab is supplied as a sterile, clear, colorless, preservative-free liquid concentrate for intravenous (IV) administration in either 100 mg (10 mL) or 500 mg (50 mL) single-use vials, which must be diluted before administration
  Standard rituximab pre-medications will be provided in preparation for the rituximab infusions.
  Other Names: Rituxan®
  Arms: Rituximab+PAH SOC
Other: Placebo — Participants receive placebo intravenous (IV) infusions 14 days apart (Day 0 and Week 2).
  Standard pre-medications will be provided in preparation for the infusions.
  Other Names: Placebo for rituximab
  Arms: Placebo + PAH SOC
Diagnostic Test: CMRI — Up to 20 participants from each treatment arm will be assessed by CMRI at Baseline and at Week 24.
  Other Names: cardiac MRI; cardiac Magnetic Resonance Imaging
Drug: prednisone — Prednisone dose of 40 mg (or equivalent) by mouth administered the night before and the morning of each study drug infusion.
  Other Names: prednisone tablets; Rayos®
Drug: methylprednisolone — Methylprednisolone (or equivalent corticosteroid) administered intravenously 30 minutes prior to each study drug infusion.
  Other Names: corticosteroid
Drug: diphenhydramine — Diphenhydramine 50 mg (or equivalent) administered by mouth approximately thirty to sixty minutes prior to each study drug infusion.
  Dose may be repeated every four hours, as needed.
  Other Names: Benadryl®
Drug: acetaminophen — Acetaminophen 650 mg (or equivalent) administered by mouth approximately thirty to sixty minutes prior to each study drug infusion.
  Dose may be repeated every four hours, as needed.
  Other Names: Tylenol®

SUMMARY:
Systemic sclerosis-associated pulmonary arterial hypertension (SSc-PAH) is a serious, life-threatening manifestation of systemic sclerosis (SSc), an autoimmune disease of the connective tissue characterized by scarring (fibrosis) and atrophy of the skin, joints and tendons, skeletal muscles, and internal organs, and immunological disturbances. One-year survival for patients with SSc-PAH ranges from 50-81%. There is currently no cure for SSc-PAH and treatment is limited to vasodilator therapy used in all forms of PAH. In recent studies, immunotherapy was shown to be effective in treating SSc-interstitial lung disease, another serious, life-threatening manifestation of SSc. In addition, there are compelling pre-clinical data and anecdotal clinical reports that suggest modulation of the immune system may be an effective strategy for treating SSc-PAH. To test this approach, this trial will determine if rituximab, an immunotherapy, has a marked beneficial effect on clinical disease progression, with minimal toxicity, in patients with SSc-PAH when compared to placebo.

DETAILED DESCRIPTION:
This prospective, double-blind, placebo-controlled, multi-center, randomized trial will evaluate the effect of rituximab on disease progression in subjects with SSc-PAH receiving concurrent stable-dose standard medical therapy with a prostanoid, endothelin receptor antagonist, and/or phosphodiesterase 5 (PDE-5) inhibitor. The study will focus on assessment of clinical response and safety measures longitudinally. In addition, the effects of treatment with rituximab on the underlying immune mechanisms associated with B-cell dysregulation and pathogenic autoantibody response in this disease will be investigated. 1000 mg of rituximab or placebo will be administered as two IV infusions given two weeks apart. Clinical assessments and sample collection will occur at monthly visits through Week 48. If a participant has not recovered B cells by Week 48, B cell studies will be conducted quarterly until reconstitution is documented or for 2 years after initial treatment.

This trial will include a sub-study, entitled "Right Ventricular Response to Rituximab in Systemic Sclerosis-Associated Pulmonary Arterial Hypertension - A Magnetic Resonance Imaging Sub-study" (RESTORE Sub-study). The objective of the RESTORE sub-study is to evaluate the therapeutic effect of rituximab on the right ventricle of patients with SSc-PAH. Changes in right ventricular end diastolic volume index (RVEDVI) and stroke volume (SV) determined by cardiac MRI will be used as surrogates of right ventricle function and prognosis. Enrollment for the RESTORE sub-study will parallel that of main trial. Twenty patients from each treatment arm, distributed among all participating sites, will be recruited for this sub-study. Each patient will be studied at baseline (i.e. prior to initiation of study drug) and after 24 weeks or at time of discontinuation. In addition to the data collection and testing specified in the main trial, participants in RESTORE will undergo comprehensive cardiac MRI evaluation. All main trial study inclusion and exclusion criteria apply, as well as additional exclusion criteria that pertain only to the RESTORE sub-study: 1) known hypersensitivity to Gadolinium; 2) inability to tolerate or cooperate with MRI; 3) morbid obesity; and 4) presence of metallic objects or pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent.
* Clinical diagnosis of systemic sclerosis (either limited or diffuse cutaneous disease).
* Diagnosis of SSc-PAH within the past 5 years, with a mean pulmonary arterial pressure of ≥ 25 mmHg at entry.
* Mean Pulmonary Vascular Resistance (PVR) of > 3 Wood units.
* Screening 6-minute Walking Distance (6MWD) of at least 100 meters.
* New York Heart Association (NYHA) Functional Class II, III, or IV.
* Subject must be able to maintain O2 saturation ≥ 90% at rest (with or without oxygen);

  --Oxygen use is permitted.
* Subject must be vaccinated with the pneumococcal vaccine at least one month prior to initiation of therapy, unless subject was vaccinated within 5 years of study entry.
* Subject must have been treated with background medical therapy for PAH (prostanoid, endothelin receptor antagonist, PDE-5 inhibitor, and/or guanylate cyclase stimulators) for a minimum of 8 weeks and have been on stable dose medical therapy for at least 4 weeks prior to randomization with no expectation of change for 24 weeks after randomization.

Exclusion Criteria:

* Documented PAH for greater than 5 years at the time of randomization defined as:

  * Measurement of a mean Pulmonary Artery Pressure (PAP) > 25 mmHg by right heart catheterization at least 5 years previously, OR
  * Treatment with targeted background PAH therapy for > 5 years.
* Pulmonary Capillary Wedge Pressure > 15 mmHg or Left Ventricular End Diastolic Pressure > 15 mmHg.
* Persistent hypotension with Systolic Blood Pressure (SBP) < 90 mmHg.
* Treatment with cyclophosphamide within 4 weeks of randomization.
* Treatment with immunocompromising biologic agents within 4 weeks prior to treatment initiation or treatment with infliximab within 8 weeks prior to treatment initiation.
* If being treated with a non-biologic immunosuppressive or immunomodulating drug, changes in dosage within 4 weeks prior to randomization. Subjects taking prednisone or equivalent corticosteroid > 10mg daily are excluded.
* Previous exposure to any lymphocyte or B cell depleting agent.
* PAH for any reason other than SSc.
* History of coronary artery disease, significant ventricular tachy-arrhythmia, stent placement, coronary artery bypass surgery, and/or myocardial infarction.
* Moderate or severe interstitial lung disease.
* Chronic infections.
* Positive serology for infection with hepatitis B or C.
* A deep space infection within the past 2 years.
* Evidence of active infection within 2 weeks of randomization
* Presence of a positive tuberculosis (TB) skin test (e.g., PPD test) or positive QuantiFERON®-TB blood test, an indeterminate QuantiFERON®-TB blood test, or latent tuberculosis (TB).
* Significant renal insufficiency.
* Active, untreated SSc renal crisis at the time of enrollment.
* Recent administration of a live vaccine (< 8 weeks) or any other immunization within 4 weeks of treatment.
* History of anaphylaxis or Immunoglobulin E (IgE) -mediated hypersensitivity to murine proteins or any component of rituximab.
* Pregnancy.
* Lactation.
* History of malignancy within the last 5 years, except for resected basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ cervical cancer Grade I.
* A woman of childbearing potential who is unwilling to use a medically acceptable form of birth control
* History of non-compliance with other medical therapies.
* History of alcohol or drug abuse within 1 year of randomization.
* Receipt of any investigational drug or device within 4 weeks before the Screening Visit, with the exception of investigational prostanoids, endothelin receptor antagonists, and PDE-5 inhibitors, and guanylate cyclase stimulators.
* Recipient of lung transplant.
* Laboratory parameters at the screening visit showing any of the following abnormal results: Transaminases > 2x the upper limit of normal (ULN) and/or bilirubin > 2x ULN; Absolute neutrophil count < 1,500/mm^3; Platelet count < 100,000/mm^3; Hemoglobin < 9 g/dL.
* Concurrent treatment in a clinical research study using a non-FDA approved agent with the exception of an open-label study/study extension of investigational prostanoids, endothelin receptor antagonists, and PDE-5 inhibitors, and guanylate cyclase stimulators, provided the open-label investigational drug will be available and dose will remain stable through the trial's primary outcome time point of 24 weeks after randomization in this study, ASC01 (NCT01086540).
* Any condition or treatment, which in the opinion of the investigator, places the subject at unacceptable risk as a participant in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-06-24 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nicolls, M.D., Study Chair — Stanford University; David B. Badesch, M.D., Study Chair — University of Colorado Health Sciences Center (Aurora, CO); Thomas A. Medsger, Jr., M.D., Study Chair — University of Pittsburgh; Lorinda Chung, MD, Study Chair — Stanford University; Robyn Domsic, MD, Study Chair — University of Pittsburgh: Division of Rheumatology and Clinical Immunology; Aryeh Fischer, MD, Study Chair — National Jewish Health: University of Colorado School of Medicine; Roham Zamanian, MD, Study Chair — Stanford University
Locations (17):
- United States (17):
  - Stanford Health Care, Stanford, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Pulmonary and Critical Care Medicine, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Health Clinics and Surgery Center, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill: UNC Hospitals, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center-William P. Clements University Hospital, Dallas, Texas
  - University of Texas: Memorial Herman Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Zamanian RT, Badesch D, Chung L, Domsic RT, Medsger T, Pinckney A, Keyes-Elstein L, D'Aveta C, Spychala M, White RJ, Hassoun PM, Torres F, Sweatt AJ, Molitor JA, Khanna D, Maecker H, Welch B, Goldmuntz E, Nicolls MR. Safety and Efficacy of B-Cell Depletion with Rituximab for the Treatment of Systemic Sclerosis-associated Pulmonary Arterial Hypertension: A Multicenter, Double-Blind, Randomized, Placebo-controlled Trial. Am J Respir Crit Care Med. 2021 Jul 15;204(2):209-221. doi: 10.1164/rccm.202009-3481OC. PMID 33651671
- [Result] Zhang Y, Michelakis ED. A Phase-2 NIH-sponsored Randomized Clinical Trial of Rituximab in Scleroderma-associated Pulmonary Arterial Hypertension Did Not Reach Significance for Its Endpoints: End of Story? Not So Fast! Am J Respir Crit Care Med. 2021 Jul 15;204(2):123-125. doi: 10.1164/rccm.202103-0612ED. No abstract available. PMID 33856964
- [Result] Andreasson K, Bengtsson MF, Bostrom C, Hesselstrand R, Volkmann ER. Multiple Manifestations of Systemic Sclerosis Affect Walk Distance. Am J Respir Crit Care Med. 2021 Aug 1;204(3):359. doi: 10.1164/rccm.202104-0938LE. No abstract available. PMID 34107236
- [Result] Zamanian RT, Pinckney A, Domsic RT, Medsger T, Keyes-Elstein L, Sweatt AJ, Welch B, Goldmuntz E, Nicolls MR, Chung L. Reply to Andreasson et al.: Multiple Manifestations of Systemic Sclerosis Affect Walk Distance. Am J Respir Crit Care Med. 2021 Aug 1;204(3):377-378. doi: 10.1164/rccm.202104-1023LE. No abstract available. PMID 34107229
- [Derived] de Bourcy CFA, Dekker CL, Davis MM, Nicolls MR, Quake SR. Dynamics of the human antibody repertoire after B cell depletion in systemic sclerosis. Sci Immunol. 2017 Sep 29;2(15):eaan8289. doi: 10.1126/sciimmunol.aan8289. PMID 28963118
- See also: The National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- See also: The Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-six study sites in the US were activated. Of these, 19 sites screened a total of 108 participants. Fifty-seven participants were randomized and study results summarized.
Groups:
- Rituximab: Rituximab (a monoclonal antibody to CD20) was administered as two IV infusions, 1000 mg each, given two weeks apart at Day 0 and Week 2. Participants were pre-treated with corticosteroids, diphenhydramine, and acetaminophen. The appearance of the packaging and solutions used to administer rituximab/placebo was identical in both study arms.
- Placebo: Placebo was administered as two IV infusions, given two weeks apart at Day 0 and Week 2. Participants were pre-treated with corticosteroids, diphenhydramine, and acetaminophen. The appearance of the packaging and solutions used to administer rituximab/placebo was identical in both study arms.
Period: Overall Study
Arm/Group | Rituximab | Placebo
Started | 29 | 28
Completed | 23 | 26
Not Completed | 6 | 2
Not completed — Death | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Addition of new therapy for PAH | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.9) | 59.1 (9.4) | 58.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 24 | 24 | 48
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 28 | 57
Six Minute Walk Test Distance (Meters) [Mean (Standard Deviation); unit: Meters] — The six minute walk test measures the distance a participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the participant to walk as far as possible in six minutes. The participant is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The total distance walked, in meters, was recorded for each participant. Longer distances indicate better outcomes.
  Meters | 338.7 (103.3) | 323.4 (97.1) | 331.2 (99.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Distance Walked During a Six Minute Walk Test
Description: The six minute walk test measures the distance a participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the participant to walk as far as possible in six minutes. The participant is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The total distance walked, in meters, was recorded for each participant. Longer distances indicate better outcomes.
Time Frame: Baseline (Pre Treatment Initiation) to Week 24
Population: The Modified Intent-to-Treat (ITT) population included all randomized participants who met entry criteria and initiated therapy. Participants who, for whatever reason, did not complete their assigned therapy were included in the ITT population in the groups to which they were randomized.
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Meters | 23.6 (11.1) | 0.5 (9.7)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; The null hypothesis was that the mean change in 6MWD between baseline and Week 24 does not differ between rituximab and placebo. A repeated measures random effect model was fit to model the distance walked as a function of treatment, visit week, a treatment by visit week interaction, and a quadratic visit term. A random slope and intercept were fit for each participant using a separate unstructured covariance matrix for each treatment group. The model included all available data up to Week 24; Test type: Superiority; p = 0.12, Mixed Models Analysis; Median Difference (Final Values) = 23.1, Standard Error of Mean 14.71 — Estimate is for the difference (Rituximab - Placebo) at Week 24

2. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance Measured by Right Heart Catheterization at Week 24
Description: During a right heart catheterization, a catheter is guided to the right side of the heart and then into the pulmonary artery; blood flow through the heart is observed and is used to measure pressures in a participant's heart and lungs. The calculation of Pulmonary Vascular Resistance (PVR) is measured in Woods Units. Change is derived by measuring the difference between Baseline and Week 24 PVR (Week 24 minus Baseline). Higher PVR values indicate worse disease status.
Time Frame: Baseline (Pre Treatment Initiation) to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Woods Units
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Woods Units | -0.5 (0.36) | 0.1 (0.61)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures mixed model was fit with PVR as the outcome and treatment, visit week (actual observed week), and their interaction as predictors. Random intercepts and slopes were fit for each participant using an unstructured covariance structure for each treatment group; Test type: Superiority; p = 0.42, Mixed Models Analysis — P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.71

3. Secondary Outcome: Change From Baseline in Distance Walked During a Six Minute Walk Test at Week 24 and Week 48
Description: as for outcome 1
Time Frame: Baseline (Pre Treatment Initiation) to Week 24 and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Meters
  Change from Baseline to Week 24 | 25.5 (8.8) | 0.4 (7.4)
  Change from Baseline to Week 48 | 9.5 (12.4) | -7.0 (8.6)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures random effect model was fit to model the distance walked as a function of treatment, visit week, a treatment by visit week interaction, and a quadratic visit term. A random slope and intercept were fit for each participant using a separate unstructured covariance matrix for each treatment group. The model included all available data up to Week 48; Test type: Superiority; p = 0.28, Mixed Models Analysis — Week 48 value. P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = 16.4, Standard Error of Mean 15.1 — Estimate is for the difference (Rituximab - Placebo) at Week 48
Statistical Analysis 2: Comparison: Rituximab vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.031, Mixed Models Analysis — Week 24 value. P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = 25.1, Standard Error of Mean 11.5 — Estimate is for the difference (Rituximab - Placebo) at Week 24

4. Secondary Outcome: Time to Clinical Worsening
Description: Assessment of time to clinical worsening, censored at Week 48, defined as the first occurrence of any of the following:
  * death,
  * hospitalization for Systemic Sclerosis-Associated Pulmonary Arterial Hypertension (SSc-PAH),
  * lung transplantation,
  * atrial septostomy,
  * addition of other Pulmonary Arterial Hypertension (PAH) therapeutic agents, or
  * worsening of the six minute walk distance by > 20% and an increase in New York Heart Association functional class.
  Time to clinical worsening was defined as the first date that met any of the above criteria and was calculated in study days as: date of first event minus (-) date of treatment randomization. If a participant did not experience any of the referenced events by Week 48 or, if the date of death was after the 48 week follow-up period, time to clinical worsening was equal to the participant's duration of follow-up in the study.
Time Frame: Baseline (Pre Treatment Initiation) to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Weeks | 21.2 (14.2) | 26.2 (4.0)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Kaplan-Meier curves for time to clinical worsening were compared using a log-rank test; Test type: Superiority; p = 0.92, Log Rank — P-values not adjusted for multiple comparisons

5. Secondary Outcome: Time to the Change or Addition of New Pulmonary Arterial Hypertension (PAH) Therapeutic Medications
Description: Per protocol, from the time of study entry, participants were to remain on background PAH medical therapy with either a single agent or a combination of prostanoid, endothelin receptor antagonist, PDE-5 inhibitor, and/or guanylate cyclase stimulators as per the entry criteria. Doses should have remained stable through the Week 24 primary outcome/endpoint visit. If a dose of a background PAH medication was changed or a new PAH medication was added during the course of the trial, the date of the first dose change or additional medication was recorded. Time to the addition or modification of PAH medications was defined in study days as: date of the first time a PAH medication was modified or added minus (-) date of randomization.
Time Frame: Baseline (Pre Treatment Initiation) to Week 48
Population: The Modified Intent-to-Treat (ITT) population included all randomized participants who met entry criteria and initiated therapy. Participants who, for whatever reason, did not complete their assigned therapy were be included in the ITT population in the groups to which they were randomized.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Weeks | 21.2 (14.4) | 26.7 (3.9)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Kaplan-Meier curves for time to change or addition of PAH medications were compared using a log-rank test; Test type: Superiority; p = 0.36, Log Rank — P-values not adjusted for multiple comparisons

6. Secondary Outcome: Change From Baseline in Quality of Life as Measured by the Short Form Health Survey (SF-36): Mental Component Summary Score
Description: The SF-36 measures health-related quality of life. It has 36 items and 2 component scores, the Physical Component Score and the Mental Component Score. The SF-36 Mental Health component summary score is comprised of the Vitality Scale, the Social Functioning Scale, the Role-Emotional Scale, and the Mental Health Scale. It is scaled from 0 to 100 with a score of 0 equivalent to maximum disability and a score of 100 is equivalent to no disability. A negative value indicates a decrease in quality of life from Baseline.
Time Frame: Baseline (Pre Treatment Initiation) to Week 24 and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Units on a Scale
  Change from Baseline to Week 24 | 0.1 (0.9) | 0.4 (1.0)
  Change from Baseline to Week 48 | 0.2 (1.8) | 0.9 (1.9)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures random effect model was fit with the mental component score as the outcome, and treatment, visit week (actual observed week), and their interaction as predictors. Random intercepts and slopes were fit for each participant using an unstructured covariance structure for each treatment group; Test type: Superiority; p = 0.81, Mixed Models Analysis — P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.6, Standard Error of Mean 2.7 — Estimate is for the difference (Rituximab - Placebo) at Week 48

7. Secondary Outcome: Change From Baseline in Quality of Life as Measured by the Short Form Health Survey (SF-36): Physical Component Summary Score
Description: The SF-36 measures health-related quality of life. It has 36 items and 2 component scores, the Physical Component Score and the Mental Component Score. The SF-36 Physical component summary score is comprised of the Physical Functioning Scale, the Role-Physical Scale, the Bodily Pain Scale, and the General Health Scale. It is scaled from 0 to 100 with a score of 0 equivalent to maximum disability and a score of 100 is equivalent to no disability. A negative value indicates a decrease in quality of life from Baseline.
Time Frame: Baseline (Pre Treatment Initiation) to Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Units on a Scale
  Change from Baseline to Week 24 | 0.6 (0.8) | 1.7 (0.7)
  Change from Baseline to Week 48 | 1.3 (1.5) | 3.5 (1.5)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures random effect model was fit with the physical component score as the outcome, and treatment, visit week (actual observed week), and their interaction as predictors. Random intercepts and slopes were fit for each participant using an unstructured covariance structure for each treatment group; Test type: Superiority; p = 0.30, Mixed Models Analysis — P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = -2.2, Standard Error of Mean 2.1 — Estimate is for the difference (Rituximab - Placebo) at Week 48

8. Secondary Outcome: Change in Quality of Life as Measured by the Disability Index of the Scleroderma Health Assessment Questionnaire (HAQ-DI)
Description: The HAQ-DI is a self-reported questionnaire of functionality that includes questions in 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities) and addresses scleroderma related manifestations that contribute to disability. The final score ranges from 0 to 3, where a higher HAQ-DI score indicates a worse outcome.
Time Frame: Baseline (Pre Treatment Initiation) to Week 24 and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Units on a Scale
  Change from Baseline to Week 24 | 0.0 (0.05) | 0.0 (0.02)
  Change from Baseline to Week 48 | 0.0 (0.09) | 0.0 (0.05)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures random effect model was fit with HAQ-DI as the outcome, and treatment, visit week (actual observed week), and their interaction as predictors. Random intercepts and slopes were fit for each participant using an unstructured covariance structure for each treatment group; Test type: Superiority; p = 0.58, Mixed Models Analysis — P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.11 — Estimate is for the difference (Rituximab - Placebo) at Week 48

9. Secondary Outcome: Number of New Digital Ulcers
Description: The total number of digital ulcers present on the dorsal and palmar surfaces for both the left and right fingers were captured at the Baseline study visit. The number of new digital ulcers since the last study visit (including any ulcers that had appeared and healed since the last study visit) on the dorsal and palmar surfaces for both the left and right fingers were captured at the post-Baseline study visits. The total number of digital ulcers on both hands was summed from the number present on the dorsal and palmar surfaces for both the left and right fingers.
Time Frame: Baseline (Pre Treatment Initiation) to Week 24 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: New Ulcers
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
New Ulcers
  Total Ulcer Count at Baseline | 0.6 (2.04) | 0.4 (1.58)
  New Ulcers at Week 24 | 0.0 (0.00) | 0.1 (0.59)
  New Ulcers at Week 48 | 0.1 (0.29) | 0.2 (0.63)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A Poisson model was used to describe the rate of new digital ulcers (per week) as the outcome with treatment, number of digital ulcers at Baseline, and if the measurement was affected by changed or new PAH therapeutic agents as covariates; Test type: Superiority; p = 0.47, Regression, Linear — P-values not adjusted for multiple comparisons

10. Secondary Outcome: Change in Severity of Raynaud's Phenomenon
Description: Severity of Raynaud's phenomenon was measured by a Visual Analog Scale (VAS) of the Scleroderma Health Assessment Questionnaire (SHAQ). The SHAQ VAS includes a question asking, "In the past week, how much has your Raynaud's Phenomenon interfered with your activities?" Participants were asked to place a mark on a 15 cm line, scaled from 0 (does not interfere) to 100 (very severe limitation), to describe the severity of their Raynaud's phenomenon in the past week. The distance from the left edge of the line to the vertical line placed by the participant was measured in centimeters; VAS scores were converted to a 0 to 100 scale.
Time Frame: Baseline (Pre Treatment Initiation) to Week 24 and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Score on a Scale
  Change from Baseline to Week 24 | -2.2 (1.8) | 0.1 (2.2)
  Change from Baseline to Week 48 | -4.4 (3.6) | 0.1 (4.4)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures random effect model was fit with severity of Raynaud's (0 to 100) as the outcome, and treatment, visit week (actual observed week), and their interaction as predictors. Random intercepts and slopes were fit for each participant using an unstructured covariance structure for each treatment group; Test type: Superiority; p = 0.43, Mixed Models Analysis — P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = -4.6, Standard Error of Mean 5.7 — Estimate is for the difference (Rituximab - Placebo) at Week 48

11. Secondary Outcome: Change in Carbon Monoxide Diffusing Capacity (DLCO)
Description: Carbon Monoxide Diffusing Capacity (DLCO) is a measure of lung function. Predicted values for DLCO were computed according to the Global Lung Function Initiative (GLI) all-age reference values and corrected for hemoglobin. Lower DLCO values indicate worse disease activity.
  DLCO (Diffusing Capacity of the Lungs for Carbon Monoxide)
Time Frame: Baseline (Pre Treatment Initiation) to Week 24 and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent Predicted Value
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Percent Predicted Value
  Change from Baseline to Week 24 | -0.3 (1.03) | 0.4 (0.95)
  Change from Baseline to Week 48 | -0.5 (2.06) | 0.7 (1.89)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures random effect model was fit with DLCO as the outcome, and treatment, visit week (actual observed week), and their interaction as predictors. Random intercepts and slopes were fit for each participant using an unstructured covariance structure for each treatment group; Test type: Superiority; p = 0.65, Mixed Models Analysis — P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = -1.3, Standard Error of Mean 2.8 — Estimate is for the difference (Rituximab - Placebo) at Week 48

12. Secondary Outcome: Oxygen Saturation Levels at Week 24 and Week 48
Description: Oxygen saturation is the amount of oxygen that is in your bloodstream and is measured as the percentage of blood hemoglobin that is carrying oxygen. Normal oxygen saturation levels are considered to be 95-100 percent; low oxygen saturation values indicate worse disease. Room air oxygen saturation by pulse oximetry and/or amount of supplemental oxygen used, if saturation <90%, were recorded.
Time Frame: Week 24 , Week 48
Population: The Modified Intent-to-Treat (ITT) population included all randomized participants who met entry criteria and initiated treatment. Participants who, for whatever reason, did not complete their assigned therapy were included in the ITT population in the groups to which they were randomized.
Measure: Mean (Standard Deviation); unit: Percent Oxygen Saturation
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Percent Oxygen Saturation
  O2 Sat Level: Week 24 | 96.5 (3.4) | 96.1 (3.9)
  O2 Sat Level: Week 48 | 97.7 (2.5) | 96.2 (4.6)

13. Secondary Outcome: Percent Change From Baseline in Pulmonary Vascular Resistance Measured by Right Heart Catheterization
Description: During a right heart catheterization, a catheter is guided to the right side of the heart and then into the pulmonary artery; blood flow through the heart is observed and is used to measure pressures in a participant's heart and lungs. Pulmonary vascular resistance (PVR) is measured in Woods Units. Higher PVR values indicate worse disease status.
  Change in PVR is determined by Baseline value minus (-) Week 24 value.
Time Frame: Baseline (Pre Treatment Initiation) to Week 24
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 27 | 27
Percent Change | -4.6 (5.5) | 3.2 (7.9)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; A repeated measures mixed model was fit with percent change in PVR as the outcome and baseline PVR, treatment, visit week (actual observed week), and their interaction as predictors. Random intercepts and slopes were fit for each participant using an unstructured covariance structure for each treatment group; Test type: Superiority; p = 0.42, Mixed Models Analysis — P-values not adjusted for multiple comparisons; Mean Difference (Final Values) = -7.9, Standard Error of Mean 9.7

14. Secondary Outcome: Number of Infusion-Related Toxicities
Description: The number of Grade 3, 4, and 5 Adverse Events (AEs), which were defined as possibly, probably, or definitely related to rituximab or placebo infusion.
  This study graded the severity of adverse events according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Day 0 (Treatment Randomization) to Week 48
Population: The Safety population included all participants for whom study treatment was initiated.
Measure: Number; unit: Events
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 29 | 28
Events
  Grade 3 AEs | 15 | 7
  Grade 4 AEs | 3 | 0
  Grade 5 AEs | 0 | 0

15. Secondary Outcome: Number of Grade 3 or Higher Adverse Events (AEs) Through Week 48
Description: Total number of Grade 3, 4, and 5 AEs. Ref: National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Baseline (Pre Treatment Initiation) to Week 48
Population: The Safety population included all participants for whom study treatment was initiated.
Measure: Number; unit: Events
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 29 | 28
Events
  Grade 3 AEs | 28 | 19
  Grade 4 AEs | 6 | 2
  Grade 5 AEs | 3 | 1

16. Secondary Outcome: Number of Infection-Related Adverse Events (AEs) Through Week 48
Description: Number of adverse events classified as infections. Reference: National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
Time Frame: Day 0 (Treatment Randomization) to Week 48
Population: The Safety population included all participants for whom study treatment was initiated.
Measure: Number; unit: Events
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 29 | 28
Events | 48 | 44

17. Secondary Outcome: Treatment-Related Mortality: From Treatment Initiation to Week 48
Description: Death occurring after randomization and ≤ Week 48, and possibly, probably, or definitely resulting from assigned study treatment.
Time Frame: Day 0 (Treatment Randomization) to Week 48
Population: The Safety population included all participants for whom study treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 29 | 28
Participants | 0 | 0

18. Secondary Outcome: All-Cause Mortality: From Treatment Initiation to Week 48
Description: Death from any cause occurring after randomization and ≤ Week 48.
Time Frame: Day 0 (Treatment Randomization) to Week 48
Population: The Safety population included all participants for whom study treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 29 | 28
Participants | 4 | 1
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Kaplan-Meier curves for time to all-cause mortality were compared using a log-rank test; Test type: Superiority; p = 0.17, Log Rank — P-values not adjusted for multiple comparisons

19. Secondary Outcome: All-Cause Mortality: From Treatment Initiation to Week 104
Description: Death from any cause occurring after randomization and ≤ Week 104.
Time Frame: Day 0 (Treatment Randomization) to Week 104
Population: The Safety population included all participants for whom study treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 29 | 28
Participants | 8 | 5
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Kaplan-Meier curves for time to all-cause mortality were compared using a log-rank test; Test type: Superiority; p = 0.35, Log Rank — P-values not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: Up to 104 weeks.
Description: AEs grade 2 and above were collected from the time the first dose of study drug/placebo until completion of study participation (to Week 48) or until 30 days after premature withdrawal (without withdrawing consent). During the quarterly monitoring for b cells period of the study (Week 48 to Week 104), only grade 3 and higher infections were collected. AEs were graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 4.0.
Arm/Group | Rituximab | Placebo
All-Cause Mortality (participants affected / at risk) | 8/29 | 5/28
Serious Adverse Events (participants affected / at risk) | 14/29 | 9/28
Other Adverse Events (participants affected / at risk) | 28/29 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=29) | Placebo (N=28)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (3) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=29) | Placebo (N=28)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 15 (17) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Nail bed infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 5 (7) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 8 (10)
Urinary tract infection (Infections and infestations) | 4 (6) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 5 (6)
Brain natriuretic peptide increased (Investigations) | 2 (2) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (6) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was powered at 50% (60 participants, 30 per arm) to detect a treatment group difference of 33 meters in the six minute walk test. Enrollment ended early with 57 participants randomized instead of the planned 60.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT01086540/Prot_001.pdf
  • Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT01086540/SAP_000.pdf